CLINICAL TRIAL: NCT01048606
Title: Exercise and Phytoestrogens: a Synergistic Effect on Factors Predisposing to CVD in Postmenopausal Women
Brief Title: Exercise and Phytoestrogens: Effect on Factors Predisposing to Cardiovascular Disease(CVD) in Postmenopausal Women
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Isabelle J Dionne, PhD, Université de Sherbrooke
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: IDionne_phyto_2008-2011
Record Dates: First submitted 2010-01-12; First posted 2010-01-13 (Estimated); Results first posted 2014-02-12 (Estimated); Last update posted 2014-02-12 (Estimated); Status verified 2013-12

CONDITIONS: Overweight
Keywords: Postmenopause; Overweight; Women; Phytoestrogens; Exercise; Cardiovascular Diseases; Risk Factors; Aging
MeSH Terms: conditions — Overweight; Motor Activity; Cardiovascular Diseases | interventions — Exercise; Phytoestrogens

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placeco + exercise (Active Comparator): Placebo (no phytoestrogen): Non-active capsules of the same size and appearance than phytoestrogens capsules will be used as a placebo (same posology, i.e. 4 caps/day) Exercise (three 1h-sessions/week)
  Interventions: Behavioral: Placebo + exercise
- Phytoestrogens without exercise (Active Comparator): Phytoestrogens (70mg/day of soy isoflavone) Without exercise (no structured exercise session)
  Interventions: Dietary Supplement: Phytoestrogens without exercise
- Phytoestrogens + exercise (Experimental): Phytoestrogens (70 mg/day soy isoflavone) Exercise (1h-sessions 3 times/week)
  Interventions: Other: Phytoestrogens + exercise
- Placebo without exercise (No Intervention): Placebo: Non-active capsules of the same size and appearance than phytoestrogens capsules will be used as a placebo (same posology, i.e. 4 caps/day) No exercise

INTERVENTIONS:
Behavioral: Placebo + exercise — Placebo: Non-active capsules of the same size and appearance than phytoestrogens capsules will be used as a placebo (same posology, i.e. 4 caps/day)
  Exercise intervention: Three weekly 1h-sessions will be held on 3 non-consecutive days. Each session comprises a total of 60 min of aerobic exercise (on an ergometer device) and resistance exercise (with elastic bands, free weights, exercise ball, etc.), and a 5-min cool down. Cues regarding exercise intensity will be offered to maintain intensity in a range of 60 to 80% of maximal heart rate (with the use of a target pulse, etc.). The exercise sessions will be led by a physical activity specialist.
  Arms: Placeco + exercise
Dietary Supplement: Phytoestrogens without exercise — Phytoestrogens: The phytoestrogen supplements will consist of 70 mg/day of soy isoflavones taken as 4 caps/day. More specifically, the daily dose of isoflavones contains 44 mg of diadzein, 16 mg of glycitein and 10 mg of genestein extracted from natural soy.
  Without exercise: participants will be asked to do only their usual activities without being involved in any kind of structured exercise sessions.
  Arms: Phytoestrogens without exercise
Other: Phytoestrogens + exercise — Phytoestrogens: The phytoestrogen supplements will consist of 70 mg/day of soy isoflavones taken as 4 caps/day. More specifically, the daily dose of isoflavones contains 44 mg of diadzein, 16 mg of glycitein and 10 mg of genestein extracted from natural soy.
  Exercise intervention: Three weekly 1h-sessions will be held on 3 non-consecutive days. Each session comprises a total of 60 min of aerobic exercise (on an ergometer device) and resistance exercise (with elastic bands, free weights, exercise ball, etc.), and a 5-min cool down. Cues regarding exercise intensity will be offered to maintain intensity in a range of 60 to 80% of maximal heart rate (with the use of a target pulse, etc.). The exercise sessions will be led by a physical activity specialist.
  Arms: Phytoestrogens + exercise

SUMMARY:
Menopause is characterized by a decrease of estrogen and progesterone levels and is associated with various changes in body composition, including an accumulation of total fat mass, a relocation of adiposity to the abdomen, deterioration of plasma lipid profile, increased risk of type 2 diabetes, and increased oxidative stress. Taken together, these changes increase the risk of developing cardiovascular disease (CVD).

Physical activity and hormone-replacement therapy (HRT) have been shown to act in synergy to improve total fat mass in postmenopausal (PM) women. Because the progesterone component of HRT has been associated with an increased CVD risk in older women with a family history of CVD, the use of HRT has become controversial. As a result, a large decrease of the use of HRT in the community has been observed and postmenopausal women (PM) have developed interest in alternative therapies. Among the possibilities, phytoestrogens have shown beneficial effects on menopausal symptoms and plasma lipids. Phytoestrogens are structurally and functionally similar to estradiol (the major estrogen in humans) but found only in plants such as soybean isoflavones. They do not exert any effect on breast cancer or/and endometrial tissue.

AIMS To examine the effects of phytoestrogens, exercise and the combination of both on lean body mass, total fat mass, visceral fat, blood lipid profile, oxidative stress markers, antioxidant system, glucose metabolism, and sex-hormone levels in obese PM women.

HYPOTHESES Women undergoing a combination of phytoestrogen treatment and an exercise program will display a greater increase in lean body mass, decrease in total and visceral fat mass, improvements in blood lipid profile, decrease in oxidative stress markers, increase in antioxidant system, improvement in glucose metabolism, and increase in sex-hormone levels than those submitted to any or one of the treatments.

A total of 120 women will be recruited. There will be 4 groups (30 women/group) undergoing exercise or not and supplemented with phytoestrogens or a placebo. The intervention is planned to last 12 mo. Key variables will be measured at baseline, and after 6 and 12 mo of intervention.

Three weekly 1h-sessions of exercise will be held on 3 non-consecutive days. The phytoestrogen supplements will consist of 70 mg/d of soy isoflavones taken as 4 caps/day.

ELIGIBILITY:
Inclusion Criteria:

* 50-70 years
* francophone or understanding French
* body mass index > 27kg/m²
* without physical disability
* without medical treatment influencing metabolism
* non smoker
* light drinker (<15 g ethanol/day = 1 alcoholic beverage)
* weight stable (< 2 kg) for 6 mo
* no participation in a supervised exercise program for 6 mo
* without HRT for at least 3 yrs
* and without menses for at least 12 mo

Exclusion Criteria:

* soy allergy
* known hepatic diseases
* asthma
* family history of accident cerebro-vascular
* personal history of a feminine cancer

Ages: 50 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2009-01; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle J Dionne, Ph.D., Principal Investigator — Université de Sherbrooke
Locations (1):
- Centre de recherche sur le vieillissement du CSSS-IUGS, Sherbrooke, Quebec, Canada

REFERENCES:
- [Background] Aubertin-Leheudre M, Lord C, Khalil A, Dionne IJ. Isoflavones and clinical cardiovascular risk factors in obese postmenopausal women: a randomized double-blind placebo-controlled trial. J Womens Health (Larchmt). 2008 Oct;17(8):1363-9. doi: 10.1089/jwh.2008.0836. PMID 18788990
- [Background] Choquette, S., D.-A. Lalancette, et al. (2009). Soy Isoflavones and Exercise: Possible Benefits for Postmenopausal Women's Cardiovascular Health. Current Women's Health Reviews 5(2): 56-62.
- [Background] Aubertin-Leheudre M, Lord C, Khalil A, Dionne IJ. Six months of isoflavone supplement increases fat-free mass in obese-sarcopenic postmenopausal women: a randomized double-blind controlled trial. Eur J Clin Nutr. 2007 Dec;61(12):1442-4. doi: 10.1038/sj.ejcn.1602695. Epub 2007 Feb 21. PMID 17311051
- [Background] Aubertin-Leheudre M, Lord C, Khalil A, Dionne IJ. Effect of 6 months of exercise and isoflavone supplementation on clinical cardiovascular risk factors in obese postmenopausal women: a randomized, double-blind study. Menopause. 2007 Jul-Aug;14(4):624-9. doi: 10.1097/gme.0b013e31802e426b. PMID 17290158
- [Result] Lebon J, Aubertin-Leheudre M, Bobeuf F, Lord C, Labonte M, Dionne IJ. Is a small muscle mass index really detrimental for insulin sensitivity in postmenopausal women of various body composition status? J Musculoskelet Neuronal Interact. 2012 Sep;12(3):116-26. PMID 22947543
- [Result] Barsalani R, Riesco E, Lavoie JM, Dionne IJ. Effect of exercise training and isoflavones on hepatic steatosis in overweight postmenopausal women. Climacteric. 2013 Feb;16(1):88-95. doi: 10.3109/13697137.2012.662251. Epub 2012 Apr 24. PMID 22530610
- [Result] Choquette S, Dion T, Brochu M, Dionne IJ. Soy isoflavones and exercise to improve physical capacity in postmenopausal women. Climacteric. 2013 Feb;16(1):70-7. doi: 10.3109/13697137.2011.643515. Epub 2012 Feb 16. PMID 22338607
- [Result] Riesco E, Choquette S, Audet M, Lebon J, Tessier D, Dionne IJ. Effect of exercise training combined with phytoestrogens on adipokines and C-reactive protein in postmenopausal women: a randomized trial. Metabolism. 2012 Feb;61(2):273-80. doi: 10.1016/j.metabol.2011.06.025. Epub 2011 Aug 23. PMID 21864865
- [Result] Riesco E, Choquette S, Audet M, Tessier D, Dionne IJ. Effect of exercise combined with phytoestrogens on quality of life in postmenopausal women. Climacteric. 2011 Oct;14(5):573-80. doi: 10.3109/13697137.2011.566652. Epub 2011 Aug 24. PMID 21864137
- [Result] Riesco E, Aubertin-Leheudre M, Maltais ML, Audet M, Dionne IJ. Synergic effect of phytoestrogens and exercise training on cardiovascular risk profile in exercise-responder postmenopausal women: a pilot study. Menopause. 2010 Sep-Oct;17(5):1035-9. doi: 10.1097/gme.0b013e3181da7915. PMID 20539245
- [Derived] Ghachem A, Marcotte-Chenard A, Tremblay D, Prud'homme D, Rabasa-Lhoret R, Riesco E, Brochu M, Dionne IJ. Obesity among postmenopausal women: what is the best anthropometric index to assess adiposity and success of weight-loss intervention? Menopause. 2021 Mar 1;28(6):678-685. doi: 10.1097/GME.0000000000001754. PMID 33651744
- [Derived] Myette-Cote E, Archambault-Therrien C, Brochu M, Dionne IJ, Riesco E. Physical fitness improvement in overweight postmenopausal women who do not lose fat mass in response to exercise training. Menopause. 2016 Oct;23(10):1122-9. doi: 10.1097/GME.0000000000000677. PMID 27326819
- [Derived] Choquette S, Riesco E, Cormier E, Dion T, Aubertin-Leheudre M, Dionne IJ. Effects of soya isoflavones and exercise on body composition and clinical risk factors of cardiovascular diseases in overweight postmenopausal women: a 6-month double-blind controlled trial. Br J Nutr. 2011 Apr;105(8):1199-209. doi: 10.1017/S0007114510004897. Epub 2010 Dec 17. PMID 21205384

RESULTS

PARTICIPANT FLOW:
Groups:
- Placeco + Exercise: Placebo (no phytoestrogen) Exercise (three 1h-sessions/week)
  Placebo + exercise: Placebo: Non-active capsules of the same size and appearance than phytoestrogens capsules will be used as a placebo (same posology, i.e. 4 caps/day)
  Exercise intervention: Three weekly 1h-sessions will be held on 3 non-consecutive days. Each session comprises a total of 60 min of aerobic exercise (on an ergometer device) and resistance exercise (with elastic bands, free weights, exercise ball, etc.), and a 5-min cool down. Cues regarding exercise intensity will be offered to maintain intensity in a range of 60 to 80% of maximal heart rate (with the use of a target pulse, etc.). The exercise sessions will be led by a physical activity specialist.
- Phytoestrogens Without Exercise: Phytoestrogens (70mg/day of soy isoflavone) Without exercise (no structured exercise session)
  Phytoestrogens without exercise: Phytoestrogens: The phytoestrogen supplements will consist of 70 mg/day of soy isoflavones taken as 4 caps/day. More specifically, the daily dose of isoflavones contains 44 mg of diadzein, 16 mg of glycitein and 10 mg of genestein extracted from natural soy.
  Without exercise: participants will be asked to do only their usual activities without being involved in any kind of structured exercise sessions.
- Phytoestrogens + Exercise: Phytoestrogens (70 mg/day soy isoflavone) Exercise (1h-sessions 3 times/week)
  Phytoestrogens + exercise: Phytoestrogens: The phytoestrogen supplements will consist of 70 mg/day of soy isoflavones taken as 4 caps/day. More specifically, the daily dose of isoflavones contains 44 mg of diadzein, 16 mg of glycitein and 10 mg of genestein extracted from natural soy.
  Exercise intervention: Three weekly 1h-sessions will be held on 3 non-consecutive days. Each session comprises a total of 60 min of aerobic exercise (on an ergometer device) and resistance exercise (with elastic bands, free weights, exercise ball, etc.), and a 5-min cool down. Cues regarding exercise intensity will be offered to maintain intensity in a range of 60 to 80% of maximal heart rate (with the use of a target pulse, etc.). The exercise sessions will be led by a physical activity specialist.
- Placebo Without Exercise: Placebo (no phytoestrogens) Without exercise (no structured exercise session) Placebo: Non-active capsules of the same size and appearance than phytoestrogens capsules will be used as a placebo (same posology, i.e. 4 caps/day).
Period: Overall Study
Arm/Group | Placeco + Exercise | Phytoestrogens Without Exercise | Phytoestrogens + Exercise | Placebo Without Exercise
Started | 28 | 15 | 26 | 10
Completed | 16 | 8 | 16 | 5
Not Completed | 12 | 7 | 10 | 5

BASELINE CHARACTERISTICS:
Population: Healthy overweight to obese postmenopausal women.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placeco + Exercise | Phytoestrogens Without Exercise | Phytoestrogens + Exercise | Placebo Without Exercise | Total
Number analyzed (Participants) | 28 | 15 | 26 | 10 | 79
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.5 (5.7) | 58.4 (4.3) | 60.5 (3.8) | 61.7 (3.9) | 60.4 (4.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 15 | 26 | 10 | 79
  Male | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Canada | 28 | 15 | 26 | 10 | 79
Body Mass Index [Mean (Standard Deviation); unit: kg/m2] | 29.8 (4.7) | 33.8 (5.8) | 30.3 (5.3) | 31.1 (2.9) | 30.9 (5.1)

OUTCOME MEASURES:

1. Primary Outcome: Body Composition: Dual-energy X-ray Absorptiometry Method
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: percent of total fat mass
Arm/Group | Placeco + Exercise | Phytoestrogens Without Exercise | Phytoestrogens + Exercise | Placebo Without Exercise
Number analyzed (Participants) | 28 | 15 | 26 | 10
percent of total fat mass | 44.5 (5.5) | 48.8 (5.0) | 43.8 (4.8) | 46.6 (2.8)

2. Primary Outcome: Plasma Lipid Profile: the Apolipoproteins (Apo-AI, Apo-AII, Apo-B), Cholesterol HDL, LDL and Triglycerides Levels Will be Determined by Clinical Analyses of Blood Sample (Obtained After 12 h Fasting State)
Time Frame: Baseline
Reporting Status: Not Posted

3. Primary Outcome: Glucose Metabolism: 2h-75g Oral Glucose Tolerance Test (OGTT) + Plasma Insulin and Glucose Concentrations (Blood Sample Analysis).
Time Frame: Baseline
Reporting Status: Not Posted

4. Primary Outcome: Markers of Oxidative Stress: Conjugated Diene Formation, Malondialdehyde, Alpha-tocopherol and Its Oxidised Form Alpha-tocopheryl Quinone. TAS Constitutes the Most Reliable Method for the Evaluation of Oxidative Stress in Vivo.
Time Frame: Baseline
Reporting Status: Not Posted

5. Primary Outcome: Quality of Life: Assessed With Questionnaires (SF-36 (General Health Perceptions), Kupperman Index, Perceived Stress Scale.
Time Frame: Baseline
Reporting Status: Not Posted

6. Primary Outcome: Plasma Fibrinogen Levels Measured With Luminescence.
Time Frame: Baseline
Reporting Status: Not Posted

7. Primary Outcome: Body Composition: Dual-energy X-ray Absorptiometry Method
Time Frame: 6 months
Reporting Status: Not Posted

8. Primary Outcome: Body Composition: Dual-energy X-ray Absorptiometry Method
Time Frame: 12 months
Reporting Status: Not Posted

9. Primary Outcome: Plasma Lipid Profile: the Apolipoproteins (Apo-AI, Apo-AII, Apo-B), Cholesterol HDL, LDL and Triglycerides Levels Will be Determined by Clinical Analyses of Blood Sample (Obtained After 12 h Fasting State)
Time Frame: 6 months
Reporting Status: Not Posted

10. Primary Outcome: Plasma Lipid Profile: the Apolipoproteins (Apo-AI, Apo-AII, Apo-B), Cholesterol HDL, LDL and Triglycerides Levels Will be Determined by Clinical Analyses of Blood Sample (Obtained After 12 h Fasting State)
Time Frame: 12 months
Reporting Status: Not Posted

11. Primary Outcome: Glucose Metabolism: 2h-75g Oral Glucose Tolerance Test (OGTT) + Plasma Insulin and Glucose Concentrations (Blood Sample Analysis).
Time Frame: 6 months
Reporting Status: Not Posted

12. Primary Outcome: Glucose Metabolism: 2h-75g Oral Glucose Tolerance Test (OGTT) + Plasma Insulin and Glucose Concentrations (Blood Sample Analysis).
Time Frame: 12 months
Reporting Status: Not Posted

13. Primary Outcome: Markers of Oxidative Stress: Conjugated Diene Formation, Malondialdehyde, Alpha-tocopherol and Its Oxidised Form Alpha-tocopheryl Quinone. TAS Constitutes the Most Reliable Method for the Evaluation of Oxidative Stress in Vivo.
Time Frame: 6 months
Reporting Status: Not Posted

14. Primary Outcome: Markers of Oxidative Stress: Conjugated Diene Formation, Malondialdehyde, Alpha-tocopherol and Its Oxidised Form Alpha-tocopheryl Quinone. TAS Constitutes the Most Reliable Method for the Evaluation of Oxidative Stress in Vivo.
Time Frame: 12 months
Reporting Status: Not Posted

15. Primary Outcome: Sex-hormone Levels. Estradiol, Estrone, Progesterone, Testosterone and SHBG Will be Obtained by Enzyme Immuno Assay (EIA)
Time Frame: Baseline
Reporting Status: Not Posted

16. Primary Outcome: Sex-hormone Levels. Estradiol, Estrone, Progesterone, Testosterone and SHBG Will be Obtained by Enzyme Immuno Assay (EIA)
Time Frame: 6 months
Reporting Status: Not Posted

17. Primary Outcome: Sex-hormone Levels. Estradiol, Estrone, Progesterone, Testosterone and SHBG Will be Obtained by Enzyme Immuno Assay (EIA)
Time Frame: 12 months
Reporting Status: Not Posted

18. Primary Outcome: Quality of Life: Assessed With Questionnaires (SF-36 (General Health Perceptions), Kupperman Index, Perceived Stress Scale
Time Frame: 6 months
Reporting Status: Not Posted

19. Primary Outcome: Quality of Life: Assessed With Questionnaires (SF-36 (General Health Perceptions), Kupperman Index, Perceived Stress Scale
Time Frame: 12 months
Reporting Status: Not Posted

20. Primary Outcome: Plasma Fibrinogen Levels Measured With Luminescence.
Time Frame: 6 months
Reporting Status: Not Posted

21. Primary Outcome: Plasma Fibrinogen Levels Measured With Luminescence.
Time Frame: 12 months
Reporting Status: Not Posted

22. Secondary Outcome: Dietary Intakes: 3-days Food Record. Dietary Analyses Will be Completed Using the Nutifiq Software (Université Laval)
Time Frame: 0, 6 and 12 months
Reporting Status: Not Posted

23. Secondary Outcome: Physical Activity Level: Physical Activity Scale for the Elderly (PASE)
Time Frame: 0, 6 and 12 months
Reporting Status: Not Posted

24. Secondary Outcome: Plasma Isoflavones (Diadzein) - a Marker of Phytoestrogen Compliance - Will be Measured by the ELISA Method
Time Frame: 0, 6 and 12 months
Reporting Status: Not Posted

25. Secondary Outcome: Metabolic Rate at Rest: During 30 Minutes With a Breathing Mask by Indirect Calorimetry (CCM/D, Medgraphics Corp, St-Paul, MN, USA) After a 12-hour Fast, in the Early Morning.
Time Frame: 0, 6 and 12 months
Reporting Status: Not Posted

26. Secondary Outcome: Maximal Oxygen Uptake Measured Using a Continuous, Incremental Protocol (Balke Modified Protocol) on a Treadmill With a Breathing Mask by Indirect Calorimetry (CCM/D, Medgraphics Corp, St-Paul, MN, USA).
Time Frame: 0 and 12 months
Reporting Status: Not Posted

27. Secondary Outcome: Physical Capacity: 3 Tests From the Senior Fitness Test (Chair Stand Test, Chair Sit-and-Reach Test, Back Scratch Test) + Handgrip Strength Test (Lafayette Hand Dynamometer, Indiana)
Time Frame: 0, 6 and 12 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse event data were collected during 12 months.
Arm/Group | Placeco + Exercise | Phytoestrogens Without Exercise | Phytoestrogens + Exercise | Placebo Without Exercise
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/15 | 0/26 | 0/10
Other Adverse Events (participants affected / at risk) | 0/28 | 0/15 | 0/26 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No